CLINICAL TRIAL: NCT03484936
Title: Safety and Efficacy of Remote Ischemic Conditioning in Patients With Spontaneous Intracerebral Hemorrhage
Acronym: SERIC-sICH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yi Yang (Other)
Responsible Party: Sponsor-Investigator, Yi Yang, Associated Dean of First Hospital of Jilin University, The First Hospital of Jilin University
Organization: The First Hospital of Jilin University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SERIC-sICH
Record Dates: First submitted 2018-03-25; First posted 2018-04-02 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-02

CONDITIONS: Intracranial Hemorrhages
Keywords: Intracranial Hemorrhages; remote ischemic conditioning
MeSH Terms: conditions — Intracranial Hemorrhages

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RIC+Standard medical treatment (Active Comparator): Remote ischemic conditioning (RIC) is induced by 4 cycles of 5 min of healthy upper limb ischemia followed by 5 min reperfusion. Limb ischemia was induced by inflations of a blood pressure cuff to 200 mm Hg. RIC will be conducted twice daily for 7 days. Additionally,the patients will be treated with standard medical treatment according to 2014 chinese guideline for the diagnosis and treatment of intracerebral hemorrhage.
  Interventions: Procedure: Remote ischemic conditioning
- Sham RIC+Standard medical treatment (Placebo Comparator): Sham remote ischemic conditioning (Sham RIC) is simulated by the measurement of blood pressure twice daily for 7 days.Additionally,the patients will be treated with standard medical treatment according to 2014 chinese guideline for the diagnosis and treatment of intracerebral hemorrhage.
  Interventions: Procedure: Sham remote ischemic conditioning

INTERVENTIONS:
Procedure: Remote ischemic conditioning — Remote ischemic conditioning (RIC) is induced by 4 cycles of 5 min of healthy upper limb ischemia followed by 5 min reperfusion. Limb ischemia was induced by inflations of a blood pressure cuff to 200 mm Hg. RIC will be conducted twice daily for 7 days.
  Other Names: RIC
  Arms: RIC+Standard medical treatment
Procedure: Sham remote ischemic conditioning — Sham remote ischemic conditioning (Sham RIC) is simulated by the measurement of blood pressure twice daily for 7 days.
  Other Names: Sham RIC
  Arms: Sham RIC+Standard medical treatment

SUMMARY:
The purpose of this study is to determine whether treatment with remote ischemic conditioning is of sufficient promise to improve outcome before conducting a larger clinical trial to examine its effectiveness as a treatment for intracerebral hemorrhage.

DETAILED DESCRIPTION:
Intracerebral hemorrhage is a devastating disease with a high rate of severe disability and death, while no specific treatment has been proven to improve functional outcome. As a result, new approaches need to be developed to treat intracerebral hemorrhage. Animal and human trials showed treatment with remote ischemic conditioning was safe for intracerebral hemorrhage. And repetitive remote ischemic conditioning has been shown to improve sensorimotor and neuropathological outcomes following experimental hemorrhagic stroke. Therefore, we hypothesize that repetitive remote ischemic conditioning could improve functional outcome in patients with intracerebral hemorrhage. We design this prospective, multicenter, randomized controlled double-blind trial to determine whether treatment with remote ischemic conditioning is of sufficient promise to improve outcome before conducting a larger clinical trial to examine its effectiveness as a treatment for intracerebral hemorrhage.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Supratentorial intracerebral hemorrhage confirmed by brain CT scan
3. Functional independence prior to ICH, defined as pre-ICH mRS ≤ 1
4. NIHSS score ≥ 4 and GCS ≥ 6 upon presentation
5. Able to commence RIC treatment within 12 hours of stroke onset
6. Signed and dated informed consent is obtained.

Exclusion Criteria:

1. Definite evidence of secondary ICH, such as structural abnormality, brain tumor, thrombolytic drug, and other causes
2. A very high likelihood that the patient will die within the next 24 hours on the basis of clinical and/or radiological criteria
3. Already booked for surgical treatment
4. Life expectancy of less than 90 days due to comorbid conditions
5. Severe hematologic disease
6. Concurrent use of anticoagulation drugs including Warfarin, dabigatran, rivaroxaban.
7. Concurrent use of glibenclamide or nicorandil
8. Any soft tissue, orthopedic, or vascular injury, wounds or fractures in healthy upper limb which may pose a contraindication for application of RIC
9. Severe hepatic and renal dysfunction
10. Platelet count <100×10^9/L
11. Coagulopathy defined as INR,APTT,and PT beyond the upper limit of normal range
12. Known pregnancy, or positive pregnancy test, or breastfeeding
13. Patients being enrolled or having been enrolled in other clinical trial within 3 months prior to this clinical trial
14. A high likelihood that the patient will not adhere to the study treatment and follow up regimen
15. Patients unsuitable for enrollment in the clinical trial according to investigators decision making.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 530 (Estimated)
Dates: Start 2026-03-15 (Estimated); Primary Completion 2026-09-15 (Estimated); Study Completion 2027-06-15 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with Modified Rankin Scale (mRS) Score 0-2 | 3 months
  The primary outcome measure of efficacy is the modified Rankin Scale (mRS) score, dichotomized to define good functional outcome as mRS 0-2 at 90 days.

SECONDARY OUTCOMES:
Frequency of adverse events | 3 months
  The safety endpoints will include all adverse events until day-7 or discharge (whichever is earlier), and severe adverse events through day-90 after the onset of intracerebral hemorrhage.

OTHER OUTCOMES:
Proportion of hematoma growth | 24 hours
  The proportional growth in hematoma volume during the first 24h after the onset of intracerebral hemorrhage.
Proportion of hematoma absorption | 14 days
  The proportional change in hematoma volume between 24h and 14 days or discharge (whichever is earlier) after the onset of intracerebral hemorrhage.
Changes of hematological indicators | 24 hours; 7 days
  The changes of hematological indicators (inflammatory cytokine,et al.) during the first 24h and 7 days after the onset of intracerebral hemorrhage.

CONTACTS AND LOCATIONS:
Overall Officials: Yi Yang, MD, PhD, Study Chair — Neuroscience Center, Department of Neurology, The First Hospital of Jilin University
Locations (1):
- First Hospital of Jilin University, Changchun, Jilin, China